CLINICAL TRIAL: NCT00161096
Title: Comparison of the Percentage Chronic on-Demand Users Treated With 20 Mg Pantoprazole on-Demand and Placebo o.d Versus Placebo on-Demand and 20 Mg Pantoprazole o.d. After Symptom Relief With 20 Mg Pantoprazole o.d.
Brief Title: On-Demand Use of Pantoprazole: Determinants for Chronic Use of Acid Suppressive Medication
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY1023/NL503
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2004-11

CONDITIONS: Chronic Use of Acid Suppressive Medication; GORD; GERD; Reflux; Peptic Ulcer
Keywords: on-demand therapy; pantoprazole; gastro-oesophageal reflux disease; proton pump inhibitor; acid suppression; intermittent
MeSH Terms: conditions — Gastroesophageal Reflux; Peptic Ulcer | interventions — Pantoprazole; Pharmaceutical Preparations

INTERVENTIONS:
Drug: pantoprazole 20 mg (drug)

SUMMARY:
The purpose of this study is to investigate several aspects of chronic use of acid suppressing medication: dependence on maintenance therapy, the possibilities for on-demand use, and predictors (patient characteristics) for daily need, for on-demand use and for termination of chronic use.

DETAILED DESCRIPTION:
2-5% of the general population is chronic user of acid suppressing medication (proton pump inhibitors, H2 receptor antagonists), mostly because of gastro-oesophageal reflux disease (GORD). Prescription data from health insurances show that the number of chronic users increases every year, which has large economic consequences.

There are indications however that on-demand and intermittent therapy can be as effective as daily use. No evidence exists regarding patients who are likely to benefit from intermittent, on-demand therapy or even termination.

In this study several aspects of chronic use of acid suppressive therapy are investigated in family practice patients.

Chronic users are transferred to pantoprazole 20 mg for 4 weeks. Patients with adequate relief of symptoms are randomized in two groups for a period of 13 weeks.

group 1: daily pantoprazole 20 mg, placebo on-demand (indicative for placebo-dependency) group 2: daily placebo, pantoprazole 20 mg on-demand (indicative for pharmacological dependency) Patients visit the research nurse at the beginning of the study and at week 4, 5, 10 and 17.

In this study we are looking for patient characteristics indicative for the dependency on acid suppressive drugs and for possibilities to reduce the dose of these drugs.

Furthermore, aspects described in "secondary outcomes" will be addressed.

ELIGIBILITY:
Inclusion Criteria:

* male and female (non-pregnant, non-lactating)out-patients between 18-75
* chronic users of acid suppressive therapy for at least 180 days over the last year

Exclusion Criteria:

* stage 3, 4 oesophagitis, Barrett's oesophagus, acute peptic ulcer
* gastric hypersecretory condition, predominantly IBS symptoms, previous gastric/oesophageal surgery, pyloric stenosis
* severe, unstable comorbidities
* alarm symptoms
* malignancies in the past 5 years
* use of NSAID, systemic glucocorticoids, Cox-2 inhibitors, acetylsalicylic acid more than 150 mg daily, drugs with pH-dependent absorption, anticholinergics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276
Dates: Start 2004-03; Study Completion 2005-09

PRIMARY OUTCOMES:
The percentage of patients taking 6 or more tablets on-demand per week (averaged from week 5-17.

SECONDARY OUTCOMES:
-mean weakly consumption of on-demand tablets
-percentage of patients in placebo group requiring less than 2 tablets pantoprazole per week
-proportion of patients with adequate relief per treatment group per week
-quality of life during double-blind phase (via SF-36 and QOLRAD for GERD symptom score)
-predictors of the primary outcome (age, sex, general medical and gastrointestinal history, Hp status, BMI, lifestyle factors, personality and psychological state)
-proportion of patients successfully changed from omeprazole to pantoprazole, or from 40 mg to 20 mg
-costs during all phases
-cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Mattijs E Numans, MD, PhD, Study Chair — Julius Center for Health Sciences and Primary Care